CLINICAL TRIAL: NCT06714292
Title: Efficacy and Safety of Fluorescent Surgical Marker Clip for Tumor Localization in Laparoscopic Colorectal Surgery for Colorectal Cancer Patients : Multi-center, Randomized, Single-blind, Prospective, Non-Inferiority Trial
Brief Title: Fluorescent Approach for Refined Endoscopic Marking With Clip Localization and Identification Procedure
Acronym: FLARECLIP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KSC-CRC-01
Record Dates: First submitted 2024-11-25; First posted 2024-12-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Colon Cancer
Keywords: tattooing; localization; colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clip group (Experimental): Patients who are underwent localization of colon lesion with fluorescent clip
  Interventions: Procedure: Endoscopic Clipping
- ICG group (Active Comparator): Patients who are underwent localization of colon lesion with ICG(indocyanine green) through tattooing method
  Interventions: Procedure: ICG injection

INTERVENTIONS:
Procedure: Endoscopic Clipping — localization of colon lesion with fluorescent clip
  Arms: Clip group
Procedure: ICG injection — localization of colon lesion with ICG(indocyanine green) through endoscopic tattooing
  Other Names: ICG tattooing
  Arms: ICG group

SUMMARY:
* Title of the Study Testing a Fluorescent Surgical Marker Clip for Tumor Localization in Minimally Invasive Colorectal Surgery
* Purpose of the Study This study aims to determine if a fluorescent surgical marker clip can accurately and safely localize tumor locations in the colon during minimally invasive colorectal surgery. The study will compare the effectiveness of this clip to the current method using a dye called Indocyanine Green (ICG).

The main questions the investigators aim to address are:

Can the clip safely and effectively localize tumor sites compared to ICG dye? What side effects or medical issues might arise with the use of the clip?

-Study Design Assignment

Participants will be randomly assigned to one of two groups:

The clip group: A fluorescent clip will be placed near the tumor. The dye group: ICG dye will be injected near the tumor.

Procedures Participants will undergo a colonoscopy to mark the tumor location before surgery using either the fluorescent clip or ICG dye.

* Follow-Up Participants will attend follow-up visits after surgery to monitor for any side effects or complications.
* Eligibility Inclusion Criteria

Participants may qualify if:

They are 19 years or older. They are scheduled for minimally invasive colorectal surgery for a tumor or suspected tumor.

Exclusion Criteria

Participants cannot enroll if:

They have certain medical conditions, such as blood clotting disorders or allergies to metals or iodine.

They are pregnant or breastfeeding.

-Participant Role By participating, individuals will contribute to advancing research aimed at improving methods for tumor localization during surgery, potentially leading to enhanced surgical outcomes in the future.

For questions or concerns, participants are encouraged to contact the investigators or the research team.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19years or more
* With colonic neoplasm planning minimally invasive surgery
* Need localization of lesion before surgery

Exclusion Criteria:

* Planned total proctocolectomy
* Contraindication of colonoscopy
* On pregnancy or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of localization | In operation
  Accuracy of Identifying the Exact Tumor Location
  Experimental Group: Considered successful when the tumor can be observed through the applied clips using fluorescence imaging.
  Control Group: Considered successful when the ICG-tattooed tumor can be observed.

SECONDARY OUTCOMES:
Reconfirmation Rate via Intraoperative Colonoscopy (%) | In operation
  The proportion of cases where intraoperative colonoscopy was performed.
Total Operation Time (minutes) | From start of operation to end of operation.
  The time from skin incision to skin closure.
Time Required for Endoscopic Marking Procedure (minutes) | From identifying of tumor in colonoscopy to completing the clipping or injection of ICG
  The time from identifying the tumor to completing the attachment of all required clips for marking the tumor or completing the injection of ICG.
Longitudinal Length of ICG Spread in the Control Group (mm) | After resection of colon, in operation
  In ICG group, measure the length of tattooed area using a disposable paper ruler on the serosa side of colon.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Won Park, M.D., Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Seoul Boramae Medical Center, Seoul